CLINICAL TRIAL: NCT01733290
Title: Botulinum Toxin Urethral Sphincter Injection for Dysfunctional Voiding - A Multicenter Study, Randomized, Double-Blind, Placebo Control
Brief Title: Botulinum Toxin Urethral Sphincter Injection for Dysfunctional Voiding
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Director of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TCGHUROL006
Record Dates: First submitted 2012-11-08; First posted 2012-11-27 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Dysfunctional Voiding
Keywords: Botulinum Toxin A (BoNT-A); Dysfunctional voiding
MeSH Terms: interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin A (Experimental): A total of 100 units of BoNT-A will be injected deeply into the external sphincter at the 3, 6, 9 and 12 o'clock positions in approximate equal aliquot.
  Interventions: Drug: Botulinum toxin A
- Control arm-Normal saline instillation (Placebo Comparator): Normal saline instillation
  Interventions: Drug: Normal saline instillation

INTERVENTIONS:
Drug: Botulinum toxin A — A total of 100 units of BoNT-A will be injected deeply into the external sphincter at the 3, 6, 9 and 12 o'clock positions in approximate equal aliquot.
  Other Names: Botulinum Toxin A (BoNT-A)
  Arms: Botulinum toxin A
Drug: Normal saline instillation — Normal saline instillation
  Other Names: N/S
  Arms: Control arm-Normal saline instillation

SUMMARY:
This study is designed and aimed at determine the clinical efficacy of BoNT-A on patients with dysfunctional voiding. The results of this study can provide further information for patient selection and therapeutic duration.

DETAILED DESCRIPTION:
This study is designed in a randomized, double-blind, placebo controlled, multicentric trial. A total of 60 patients will be enrolled. All patients have suffered from dysfunctional voiding that is refractory to conventional treatment. The enrolled patients should have severe dysuria or urinary retention, large residual urine and have been treated with medication or other therapeutic modality for over 3 months. The patients will be randomly assigned to allocate in the treatment and control groups in a 2:1 ratio. About 40 and 20 patients will be enrolled in the treatment and control group, respectively.

This study should be approved by the Institutional Review Board (IRB) and ethical committee of the hospital. Every patient should be thoroughly informed and written informed consent should be obtained before treatment.

Patients will receive a complete urological work-up before treatment, including urinalysis, urine culture, cystoscopy to prove no anatomical stricture or lower urinary tract pathology, and videourodynamic study. All medication that may affect the lower urinary tract function will be stopped at least 1 week before Botulinum Toxin A (BoNT-A) injection.

Videourodynamic study will be performed with the patient in supine position if patients cannot stand up or sit on the commode. A 6 Fr dual channel urethral pressure profiles (UPP) urethral catheter will be inserted to the urinary bladder. After evacuation of the residual urine, urethral pressure profilometry will be performed first. Then the bladder will be filled with normal saline containing 20% urografin at the filling rate of 30 ml/min. The filling and voiding cystourethrography will be investigated by a C-arm positioned below the patient. Uroflowmetry is recorded by a weighed transducer placed below the examination table. After the bladder is filled to the capacity, the patients are asked to urinate per urethrae. If patient cannot urinate per urethrae with the urethral catheter in situ, suprapubic puncture with a 18 Gauge needle and a 3-Fr epidural catheter will be undertaken and patients will urinate without the catheter in the urethra. The patients are requested to stand up and urinate into the commode. Pressure flow study and concomitant voiding cystourethrography are performed.

The urodynamic parameters include maximal urethral closure pressure (MUCP), functional profile length (FPL), cystometric bladder capacity (CBC), bladder compliance, voiding detrusor pressure (Pdet), maximal flow rate (Qmax), voided volume, and postvoid residual urine volume (PVR). In the patients who have detrusor underactivity, the abdominal pressure to urinate and the detrusor leak point pressure will be measured. Images of voiding cystourethrography will be emphasized on the bladder neck opening, urethral sphincter relaxation, and dilatation of posterior urethra during voiding.

Patients will be admitted and BoNT-A (treatment group) or normal saline (control group) injections will be performed in the operation room where complete cardiovascular monitoring is available during the operation. BoNT-A injections are made under cystoscopy guide in male patients and injecting periurethrally in female patients. The BoNT-A will be purchased from Allergan Company (Botox, 100 units/vial, Irvine, California, U.S.A.). Each vial of BoNT-A will be diluted to 5 ml by normal saline. A total of 100 units of BoNT-A will be injected deeply into the external sphincter at the 3, 6, 9 and 12 o'clock positions in approximate equal aliquot. After BoNT-A injections, a 14 Fr Foley catheter will be indwelled routinely for 1 day and then removed. Patients will be followed up for their voiding conditions. When dysuria persists, intermittent catheterization will be advised instead of indwelling Foley catheter. Antibiotics will not be necessary unless urinary tract infection occurs, and medications to reduce urethral sphincteric resistance are discontinued.

Patients will be closely contacted and monitored by the research assistant by telephone. They will be followed up at out-patient clinic at 1 week, 2 weeks and 4 weeks after BoNT-A injections. After the first month after initial BoNT-A injection, patients will be followed up monthly until the therapeutic effect is gone. Videourodynamic study and UPP study will be performed at 4 weeks after BoNT-A injections. The subjective improvement of voiding condition will be assessed by the obstructive symptom scores (including hesitancy, intermittency, dysuria, small caliber of urine) and quality of life score which are adopted from the International Prostate Symptom Score (IPSS) system.

The primary end-point is the change of Patient Perception of Bladder Condition (PPBC) at 4 weeks after the initial injection. If patients have a PPBC improved by two scales, they are considered as successfully treated, otherwise failed treatment. The subjective symptom score, quality of life score and urodynamic parameters will be compared at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups. For the patients who do not have significant improvement 4 weeks after BoNT-A injections, a second injection with 100 units of BoNT-A will be performed at 4 weeks after the initial injection regardless the patient's initial grouping. These patients will be followed up at the same interval until the return of voiding dysfunction.

Continuous variables are presented as means ± standard deviations (SDs), and categorical data are presented as numbers and percentages (%). Statistical comparisons within group will be performed by paired t test, between the groups are tested using the chi-square test for categorical variables, and the Wilcoxon rank-sum test for continuous variables. Long-term successful results are compared using Kaplan-Meier analyses. Statistical assessments are considered significant when p < 0.05. Statistical analyses will be performed using SPSS 15.0 statistical software (SPSS Inc., Chicago, IL).

Any side effect related to the BoNT-A injections will be asked to report. There has not been reported to have serious side effect from local injection of BoNT-A to the urethral sphincter. However, the potential side effects, such as exacerbation of urinary incontinence, allergy and anaphylactic shock should be informed to the patients and carefully monitor the postoperative conditions. Urinalysis will be checked at the first follow-up 1 and 2 week after BoNT-A injection. Antibiotics will be given if patients have significant urinary tract infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults with age of 20 years old or above.
* Free of active urinary tract infection.
* Free of bladder outlet obstruction on enrollment.
* Patients should have severe dysuria or urinary retention, large residual urine and have been treated with medication or other therapeutic modality for over 3 months.

Exclusion Criteria:

* Patients with severe cardiopulmonary disease and such as congestive heart failure, arrhythmia, poorly controlled hypertension, not able to receive regular follow-up.
* Patients with bladder outlet obstruction on enrollment.
* Patients with uncontrolled confirmed diagnosis of acute urinary tract infection.
* Patients have laboratory abnormalities at screening including: Alanine aminotransferase (ALT) > 3 x upper limit of normal range aspartate aminotransferase (AST) > 3 x upper limit of normal range.
* Patients have abnormal serum creatinine level > 2 x upper limit of normal range.
* Patients with any contraindication to be urethral catheterization during treatment.
* Female patients who is pregnant, lactating, or with child-bearing potential without contraception.
* Patients with any other serious disease considered by the investigator not suitable for general anesthesia or in the condition to enter the trial.
* Patients participated investigational drug trial within 1 month before entering this study.
* Written informed consent has been obtained.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Net change of Patient Perception of Bladder Condition (PPBC) | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of Patient Perception of Bladder Condition (PPBC) at baseline and 4 weeks after the initial injection. If patients have a PPBC improved by two scales, they are considered as successfully treated, otherwise failed treatment.
  Safety:
  Systemic adverse events

SECONDARY OUTCOMES:
Net change of the quality of life score | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of the quality of life score at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups. Quality of life score which are adopted from the International Prostate Symptom Score (IPSS) system.
  Safety:
  Systemic adverse events
Net change of the maximal urethral closure pressure (MUCP) | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of the maximal urethral closure pressure (MUCP) at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the functional profile length (FPL) | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of the functional profile length (FPL) at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the cystometric bladder capacity (CBC) | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of cystometric bladder capacity (CBC) at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the bladder compliance | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of the bladder compliance at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the voiding detrusor pressure (Pdet) | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of the voiding detrusor pressure (Pdet) at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the maximal flow rate (Qmax) | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of the maximal flow rate (Qmax) at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the voided volume | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of the voided volume at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events
Net change of the postvoid residual urine volume (PVR) | Baseline and 4 weeks
  Efficacy:
  Efficacy measured the net change of the residual urine volume (PVR) at baseline and 4 weeks after BoNT-A injection within and between the treatment group and control groups.
  Safety:
  Systemic adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital and Tzu Chi University
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

REFERENCES:
- [Background] Blaivas JG. Pathophysiology of lower urinary tract dysfunction. Urol Clin North Am. 1985 May;12(2):215-24. PMID 4039484
- [Background] Elbadawi A, Schenk EA. A new theory of the innervation of bladder musculature. 4. Innervation of the vesicourethral junction and external urethral sphincter. J Urol. 1974 May;111(5):613-5. doi: 10.1016/s0022-5347(17)60028-4. No abstract available. PMID 4856786
- [Background] Kuo HC. Effectiveness of baclofen plus terazosin treatment in patients with lower urinary tract symptoms caused by spastic urethral sphincter. Tzu Chi Med J 12:141-148, 2000.
- [Background] Kaplan SA, Ikeguchi EF, Santarosa RP, D'Alisera PM, Hendricks J, Te AE, Miller MI. Etiology of voiding dysfunction in men less than 50 years of age. Urology. 1996 Jun;47(6):836-9. doi: 10.1016/S0090-4295(96)00038-6. PMID 8677573
- [Background] Kvirkvelia L. Neocortical theta activity during learning in cats [proceedings]. Act Nerv Super (Praha). 1977 Mar;19(1):40-1. No abstract available. PMID 899636
- [Background] Carson CC, Segura JW, Osborne DM. Evaluation and treatment of the female urethral syndrome. J Urol. 1980 Nov;124(5):609-10. doi: 10.1016/s0022-5347(17)55578-0. PMID 7452783
- [Background] Raz S, Smith RB. External sphincter spasticity syndrome in female patients. J Urol. 1976 Apr;115(4):443-6. doi: 10.1016/s0022-5347(17)59235-6. PMID 944276
- [Background] Deindl FM, Vodusek DB, Bischoff C, Hofmann R, Hartung R. Dysfunctional voiding in women: which muscles are responsible? Br J Urol. 1998 Dec;82(6):814-9. doi: 10.1046/j.1464-410x.1998.00866.x. PMID 9883217
- [Background] Nitti VW, Fiske J. Cystometrogram versus cystometrogram plus voiding pressure-flow studies in women with lower urinary tract symptoms. J Urol 161(Suppl):201,1999.
- [Background] Kuo HC. Videourodynamic evaluation of the pathophysiology of lower urinary tract symptoms in neurologically intact women. Tzu Chi Med J 11:203-213,1999.
- [Background] Hinman F Jr. Nonneurogenic neurogenic bladder (the Hinman syndrome)--15 years later. J Urol. 1986 Oct;136(4):769-77. doi: 10.1016/s0022-5347(17)45077-4. PMID 3761428
- [Background] Kaplan WE, Firlit CF, Schoenberg HW. The female urethral syndrome: external sphincter spasm as etiology. J Urol. 1980 Jul;124(1):48-9. doi: 10.1016/s0022-5347(17)55287-8. PMID 7411719
- [Background] McGuire EJ, Savastano JA. Urodynamic studies in enuresis and the nonneurogenic neurogenic bladder. J Urol. 1984 Aug;132(2):299-302. doi: 10.1016/s0022-5347(17)49603-0. PMID 6737581
- [Background] Fantl JA. Behavioral intervention for community-dwelling individuals with urinary incontinence. Urology. 1998 Feb;51(2A Suppl):30-4. doi: 10.1016/s0090-4295(98)90006-1. PMID 9495733
- [Background] Carlson KV, Rome S, Nitti VW. Dysfunctional voiding in women. J Urol. 2001 Jan;165(1):143-7; discussion 147-8. doi: 10.1097/00005392-200101000-00035. PMID 11125384
- [Background] De Paepe H, Hoebeke P, Renson C, Van Laecke E, Raes A, Van Hoecke E, Van Daele J, Vande Walle J. Pelvic-floor therapy in girls with recurrent urinary tract infections and dysfunctional voiding. Br J Urol. 1998 May;81 Suppl 3:109-13. doi: 10.1046/j.1464-410x.1998.00021.x. PMID 9634033
- [Background] Wennergren H, Oberg B. Pelvic floor exercises for children: a method of treating dysfunctional voiding. Br J Urol. 1995 Jul;76(1):9-15. doi: 10.1111/j.1464-410x.1995.tb07823.x. PMID 7648068
- [Background] Vijverberg MA, Elzinga-Plomp A, Messer AP, van Gool JD, de Jong TP. Bladder rehabilitation, the effect of a cognitive training programme on urge incontinence. Eur Urol. 1997;31(1):68-72. doi: 10.1159/000474421. PMID 9032538
- [Background] Grazko MA, Polo KB, Jabbari B. Botulinum toxin A for spasticity, muscle spasms, and rigidity. Neurology. 1995 Apr;45(4):712-7. doi: 10.1212/wnl.45.4.712. PMID 7723960
- [Background] Jankovic J, Schwartz K, Donovan DT. Botulinum toxin treatment of cranial-cervical dystonia, spasmodic dysphonia, other focal dystonias and hemifacial spasm. J Neurol Neurosurg Psychiatry. 1990 Aug;53(8):633-9. doi: 10.1136/jnnp.53.8.633. PMID 2213039
- [Background] Dykstra DD, Sidi AA. Treatment of detrusor-sphincter dyssynergia with botulinum A toxin: a double-blind study. Arch Phys Med Rehabil. 1990 Jan;71(1):24-6. PMID 2297305
- [Background] Schurch B, Hauri D, Rodic B, Curt A, Meyer M, Rossier AB. Botulinum-A toxin as a treatment of detrusor-sphincter dyssynergia: a prospective study in 24 spinal cord injury patients. J Urol. 1996 Mar;155(3):1023-9. doi: 10.1016/s0022-5347(01)66376-6. PMID 8583552
- [Background] Gallien P, Robineau S, Verin M, Le Bot MP, Nicolas B, Brissot R. Treatment of detrusor sphincter dyssynergia by transperineal injection of botulinum toxin. Arch Phys Med Rehabil. 1998 Jun;79(6):715-7. doi: 10.1016/s0003-9993(98)90050-8. PMID 9630155
- [Background] Borodic GE, Joseph M, Fay L, Cozzolino D, Ferrante RJ. Botulinum A toxin for the treatment of spasmodic torticollis: dysphagia and regional toxin spread. Head Neck. 1990 Sep-Oct;12(5):392-9. doi: 10.1002/hed.2880120504. PMID 2211099
- [Background] Phelan MW, Franks M, Somogyi GT, Yokoyama T, Fraser MO, Lavelle JP, Yoshimura N, Chancellor MB. Botulinum toxin urethral sphincter injection to restore bladder emptying in men and women with voiding dysfunction. J Urol. 2001 Apr;165(4):1107-10. PMID 11257648
- [Background] Schurch B, Stohrer M, Kramer G, Schmid DM, Gaul G, Hauri D. Botulinum-A toxin for treating detrusor hyperreflexia in spinal cord injured patients: a new alternative to anticholinergic drugs? Preliminary results. J Urol. 2000 Sep;164(3 Pt 1):692-7. doi: 10.1097/00005392-200009010-00018. PMID 10953127
- [Background] Steinhardt GF, Naseer S, Cruz OA. Botulinum toxin: novel treatment for dramatic urethral dilatation associated with dysfunctional voiding. J Urol. 1997 Jul;158(1):190-1. doi: 10.1097/00005392-199707000-00067. No abstract available. PMID 9186356
- [Background] Maria G, Destito A, Lacquaniti S, Bentivoglio AR, Brisinda G, Albanese A. Relief by botulinum toxin of voiding dysfunction due to prostatitis. Lancet. 1998 Aug 22;352(9128):625. doi: 10.1016/S0140-6736(05)79580-5. No abstract available. PMID 9746032